CLINICAL TRIAL: NCT00846131
Title: A Single-Center Proof of Concept Pilot Study to Evaluate the Safety, Efficacy, and Tolerability of Sorafenib Combined With Therasphere in Subjects With Hepatocellular Carcinoma Awaiting Liver Transplantation.
Brief Title: Y-90 Alone or With Sorafenib for Pre-Transplant Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura Kulik, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU08I4; STU00005761 (Other: Northwestern University IRB)
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Subjects with primary hepatocellular carcinoma, intended for liver transplantation.
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Yttrium-90

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Y-90 alone (Active Comparator): Patients randomized to Arm A will proceed to Y-90 treatment alone in the Northwestern standard of care procedure
  Interventions: Drug: Yttrium-90 (Y-90)
- B: Sorafenib + Y-90 (Experimental): Patients randomized to Arm B will start sorafenib at a dose of 400 mg twice daily for bilirubin ≤ 1.5 x ULN and 200 mg twice daily for bilirubin > 1.5 x ULN to ≤ 3 x ULN. After 14 days of sorafenib therapy (+/- 3 days) patients will proceed to Y-90 in the Northwestern standard of care procedure
  Interventions: Drug: Sorafenib; Drug: Yttrium-90 (Y-90)

INTERVENTIONS:
Drug: Sorafenib — Randomized to Y-90 ± Sorafenib
  Other Names: BAY 54-9085 is the tosylate salt of BAY 43-9006; NEXAVAR®
  Arms: B: Sorafenib + Y-90
Drug: Yttrium-90 (Y-90) — Patients undergo radioembolization with Yttrium 90 microspheres by hepatic artery infusion
  Other Names: Radioembolization; Therasphere

SUMMARY:
A research study to determine the safety, efficacy, and tolerability of Therasphere® (also known as Y-90, or Y-90 Therasphere) combined with or without sorafenib (Nexavar®), in patients with hepatocellular carcinoma (HCC, or liver cancer), awaiting liver transplantation.

DETAILED DESCRIPTION:
Because Hepatocellular carcinoma (HCC) grows by forming new blood vessels liver transplant (OLT) offers the best chance for long term survival. However, with the growing number of patients who require OLT, prolonged wait list times often lead to drop out from the transplant list due to tumor progression. Some patients are granted an "upgrade",within the generally accepted guidelines for transplant eligibility, in order to expedite the access of patients with early HCC to transplantation before tumor progression. The use of therapies like radioembolization also known as Yttrium-90 ([Y-90] a procedure where very small beads coated with radiation are injected directly into the tumor through an artery in your groin) while awaiting OLT has become common at most transplant centers, including Northwestern, to help patients reach transplant. Additionally, these treatments are being used to move patients to a status eligible for transplant. We are studying whether a combination approach with systemic therapy and therapy applied directly to the liver, will be more successful than a single therapy . Angiogenesis (a process involving the growth of new blood vessels from pre-existing vessels) plays an important role in the early stages of HCC. A decrease in angiogenesis both locally within the treated tumor as well as in any existing tumor cells, not yet detected, would hopefully decrease the incidence of post transplant recurrence of HCC. All subjects enrolled in this study will be treated with the use of Therasphere, Y-90, which is composed of nonbiodegradable glass microspheres coated with the radioactive compound Y-90 which are injected into the hepatic artery. The concentrated radioactive microspheres within the tumor lead to "inside-out" radiation. Half of the subjects will be treated with sorafenib (NEXAVAR®) in conjunction with Y-90. The determination of which subjects will receive sorafenib will be made randomly, like the flip of a coin. Sorafenib works by slowing the growth of the tumor cell , attacking the tumor from the outside. Researchers hope to determine whether the subjects treated with sorafenib have an overall improved response to liver directed therapy with Y-90 Therasphere.

ELIGIBILITY:
Inclusion Criteria:

* Adult > 18 years olf of either gender
* Diagnosis of HCC confirmed by biopsy, CT, or MRI
* Able to carry out activities of daily living, awake >50% of waking hours
* Meets eligibility for liver transplantation
* No prior treatment for HCC
* Ability to understand and sign the informed consent
* Child-bearing women and any men agree to use two forms of birth control (one of which should be a barrier method) during the course of therapy and for 8 weeks afterward.

Exclusion Criteria:

* Less than or = 18 years old
* Ineligible for transplant due to comorbid disease
* Renal Failure requiring dialysis of any kind
* Severe Cardiac disease
* History of a stroke
* Evidence of metastatic disease- or tumors that have spread outside the liver
* Known human immunodeficiency virus (HIV) infection
* Uncontrolled blood pressure (systolic > 160) despite medication(s)
* Major surgery within 4 weeks prior to the screening visit
* Active clinically serious infection
* Serious non-healing wound, ulcer, or bone fracture.
* History of gastrointestinal bleeding (GIB) within 6 weeks prior to the screening visit
* Prior transplant of any kind
* Must be able to swallow oral pills, tablets or capsules of any size
* Use of St. John's Wort or rifampin (rifampicin).
* Currently being treated with Interferon and/or Ribavirin therapy due to the thrombocytopenias, lymphopenias and anemias observed with use of these two medications.
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any malabsorption problem
* Pregnancy or lactation. Women of childbearing potential must have a negative pregnancy test 7 days prior to beginning therapy.
* No potential living donor transplant (LDT-donor identified and worked up by the time of randomization into this study. If a living donor is later identified- the subject will be allowed to continue in the study. Sorafenib will be stopped at a minimum of 7 days prior to transplant surgery.
* Active alcohol use, drug use, or a psychiatric disease that would, in the opinion of the PI or a subinvestigator (sub-I), prevent the subject from complying with the study protocol and/or endanger the subject during their participation in the study
* Inability of the potential subject to read, understand and sign the informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2015-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To Evaluate sorafenib as an adjunct to Y-90 for control of HCC as a bridge/downstage to transplant | Up to one year
  Subjects randomized to receive Sorafenib take the drug for 2 weeks before treatment with Y90. They have imaging (CT/MRI) 2 weeks after starting Sorafenib then are treated. Post-treatment patients have blood drawn and adverse event evaluation at 2 weeks, 4 weeks, 6 weeks, and then every 6 weeks up to 1 year or time of transplant. Repeat imaging is done at 4 weeks, and then every 3 months post-treatment. Subjects not receiving Sorafenib are treated with Y90 and then are evaluated post-treatment the same as the subjects that receive the drug.

SECONDARY OUTCOMES:
To characterize the toxicity profile of sorafenib and Y90 using NCI CTC toxicity grading scales. | up to 1 year
  Subjects randomized to receive Sorafenib take the drug for 2 weeks before treatment with Y90. They have imaging (CT/MRI) 2 weeks after starting Sorafenib then are treated. Post-treatment patients have blood drawn and adverse event evaluation at 2 weeks, 4 weeks, 6 weeks, and then every 6 weeks up to 1 year or time of transplant. Repeat imaging is done at 4 weeks, and then every 3 months post-treatment. Subjects not receiving Sorafenib are treated with Y90 and then are evaluated post-treatment the same as the subjects that receive the drug.
To identify predictive and prognostic markers of how the liver cancer will respond to treatment. | up to 1 year
  All subjects are evaluated with lab work and adverse event assessment at 2, 4, and 6 weeks post-treatment, and then every 6 weeks up to 1 year or when they receive transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kulik, MD, Principal Investigator — Northwestern University, Northwestern Memorial Hospital, Northwestern Medical Faculty Foundation; Riad Salem, MD, Principal Investigator — Northwestern University, Northwestern Memorial Hospital, Northwestern Medical Faculty Foundation
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Result] Kulik L, Vouche M, Koppe S, Lewandowski RJ, Mulcahy MF, Ganger D, Habib A, Karp J, Al-Saden P, Lacouture M, Cotliar J, Abecassis M, Baker T, Salem R. Prospective randomized pilot study of Y90+/-sorafenib as bridge to transplantation in hepatocellular carcinoma. J Hepatol. 2014 Aug;61(2):309-17. doi: 10.1016/j.jhep.2014.03.023. Epub 2014 Mar 27. PMID 24681342
- [Result] Vouche M, Kulik L, Atassi R, Memon K, Hickey R, Ganger D, Miller FH, Yaghmai V, Abecassis M, Baker T, Mulcahy M, Nayar R, Lewandowski RJ, Salem R. Radiological-pathological analysis of WHO, RECIST, EASL, mRECIST and DWI: Imaging analysis from a prospective randomized trial of Y90 +/- sorafenib. Hepatology. 2013 Nov;58(5):1655-66. doi: 10.1002/hep.26487. Epub 2013 Oct 1. PMID 23703789